CLINICAL TRIAL: NCT07112742
Title: Evaluation of Short and Mid Term Effects of High Intensity Laser Therapy and Exercise in Thumb Osteoarthritis
Brief Title: Evaluation of the Effects of High Intensity Laser Therapy and Exercise in Hand Thumb Osteoarthritis
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Gizem Cengiz, Associate Professor, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025/210
Record Dates: First submitted 2025-08-01; First posted 2025-08-08 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-08

CONDITIONS: Thumb Osteoarthritis; Hand Osteoarthritis
Keywords: High Intesity Laser Therapy; Exercise; Hand Osteoarthritis; First Carpometacarpal Osteoarthritis
MeSH Terms: conditions — Motor Activity | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-Intensity Laser Therapy and Exercise (Experimental): High-intensity laser therapy will be applied to the painful and affected joint of the participants. A Class IV high-intensity laser device will be used. The parameters to be applied have been determined based on the relevant guidelines: average power 3 W, in analgesic mode, wavelength of 1064 nm, frequency of 2 Hz, energy dose of 75 J per session, spot size of 5 cm², and treatment will be administered three times per week for a total of 4 weeks. The total treatment duration will be 160 seconds. A standard exercise program including range of motion, stretching, and strengthening exercises will be administered to the participant during the treatment sessions. Strengthening exercises will be performed using a therapy ball to improve grip and pinch strength.
  Interventions: Device: High-Intensity Laser Therapy and Exercise
- High-Intensity Laser Therapy at a Non-Therapeutic Dose Combined With Exercise (Active Comparator): Participants will receive high-intensity laser therapy at an ineffective dose to the painful and affected joint. The same device as in the intervention group will be used. Due to the absence of a placebo mode in the laser device used in hospital, the lowest possible parameters will be applied to simulate an ineffective dose. For the ineffective dose, the device parameters will be set as follows: average power 0.5 W, in analgesic mode, wavelength of 1064 nm, frequency of 1 Hz, energy dose of 12 J per session, spot size of 5 cm², and treatment will be administered three times per week for a total of 4 weeks. The treatment duration will be the same as that of the intervention group. A standard exercise program including range of motion, stretching, and strengthening exercises will be administered to the participant during the treatment sessions. Strengthening exercises will be performed using a therapy ball to improve grip and pinch strength.
  Interventions: Device: High-Intensity Laser Therapy at a Non-Therapeutic Dose Combined With Exercise

INTERVENTIONS:
Device: High-Intensity Laser Therapy and Exercise — High-intensity laser therapy will be applied to the painful and affected joint of the participants. A Class IV high-intensity laser device will be used. The parameters to be applied have been determined based on the relevant guidelines: average power 3 W, in analgesic mode, wavelength of 1064 nm, frequency of 2 Hz, energy dose of 75 J per session, spot size of 5 cm², and treatment will be administered three times per week for a total of 4 weeks. The total treatment duration will be 160 seconds. A standard exercise program including range of motion, stretching, and strengthening exercises will be administered to the participant during the treatment sessions. Strengthening exercises will be performed using a therapy ball to improve grip and pinch strength.
  Arms: High-Intensity Laser Therapy and Exercise
Device: High-Intensity Laser Therapy at a Non-Therapeutic Dose Combined With Exercise — Participants will receive high-intensity laser therapy at an ineffective dose to the painful and affected joint. Due to the absence of a placebo mode in the laser device used in hospital, the lowest possible parameters will be applied to simulate an ineffective dose. For the ineffective dose, the device parameters will be set as follows: average power 0.5 W, in analgesic mode, wavelength of 1064 nm, frequency of 1 Hz, energy dose of 12 J per session, spot size of 5 cm², and treatment will be administered three times per week for a total of 4 weeks. The treatment duration will be the same as that of the intervention group. A standard exercise program including range of motion, stretching, and strengthening exercises will be administered to the participant during the treatment sessions. Strengthening exercises will be performed using a therapy ball to improve grip and pinch strength.
  Arms: High-Intensity Laser Therapy at a Non-Therapeutic Dose Combined With Exercise

SUMMARY:
One of the standard treatment methods in individuals with thumb osteoarthritis (OA) is exercise. Combination therapy options involving these exercises can be applied to patients. It has been demonstrated that high-intensity laser therapy is effective in terms of pain and function in patients with thumb OA.

The aim of this study is to investigate the effects of an exercise program combined with high-intensity laser therapy on pain, function, and muscle strength in patients with first carpometacarpal (CMC) joint osteoarthritis.

DETAILED DESCRIPTION:
First carpometacarpal (CMC) joint osteoarthritis (OA) is a common degenerative disease of the hand that causes severe pain, stiffness, weakness, and increased functional loss. It is based on joint degeneration involving articular surface deterioration, osteophyte formation, and ligamentous laxity. It is a prevalent condition in the aging population and can significantly affect hand function. The disease affects approximately 7% of men and 15% of women over the age of 50. First CMC joint OA can lead to pain and deformity at the base of the thumb, resulting in limitations in activities of daily living. Consequently, in the chronic stages of the disease, patients may experience decreased neuromuscular control of the joint, subluxation of the thumb, and adduction contracture.

The primary goals in the treatment of first CMC joint OA are to reduce pain and stiffness by improving hand function and functional capacity. Accordingly, patients are often referred to rehabilitation programs that include occupational and physical therapy interventions. High-quality studies on the conservative management of first CMC joint OA are limited. The current literature suggests that orthotic applications and intra-articular hyaluronate or steroid injections provide only partial therapeutic effects. Exercise therapy combined with patient education has been reported to be effective in the management of hand OA. Recent reviews indicate that therapeutic exercises combined with manual therapy and orthotic use may be effective in reducing pain and improving function in the short term in first CMC joint OA.

Laser therapy is a non-invasive treatment method that, through its photobiomodulation effect on cells and tissues, helps increase the rate of healing and supports tissue repair, while also reducing inflammation and alleviating pain. Although low-level laser therapy has been studied in individuals with first CMC joint OA and shown to be effective on grip strength, it has not been found to be more effective than placebo in terms of pain reduction. In another study, high-intensity laser therapy applied alone to the first CMC joint showed short-term effects on pain, but its effectiveness decreased in follow-up assessments. A study on knee osteoarthritis demonstrated that an exercise program combined with high-intensity laser therapy was more beneficial.

The hypothesis of this study is that combining high-intensity laser therapy with exercise therapy will be more effective in reducing pain over the long term in patients with first CMC joint OA.

Exercise programs have no known side effects. Possible side effects of laser therapy include erythema, hypoesthesia, hyperesthesia, petechiae, and thermal hypersensitivity. Detailed descriptions of the exercise protocol, high-intensity laser therapy protocol, and references are provided in the research protocols.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with stage I, II, or III carpometacarpal joint osteoarthritis in their dominant hand based on radiographic findings according to the Eaton-Littler-Burton classification system
* Patients experiencing pain equal to or greater than 4 on the Visual Analog Scale during activities of daily living
* Patients who agree to complete the provided clinical evaluation scales to assess treatment efficacy and who can sign the informed consent form

Exclusion Criteria:

* Patients with a history of neurological diseases affecting the upper extremity
* Patients with a history of rheumatological diseases
* Patients who have received any treatment for hand problems (including intra-articular joint injections) within the last six months
* Patients with severe hand and wrist injuries (such as fractures)
* Patients with a surgical history related to the thumb
* Patients diagnosed with hand or finger tenosynovitis, Dupuytren's disease, or Carpal Tunnel Syndrome
* Patients with conditions contraindicating laser therapy (cardiac pacemaker, cancer, pregnancy, uncontrolled diabetes mellitus, uncontrolled hypertension)

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | Patients will be assessed before and after the intervention, and at the 1st and 3rd months following the treatment.
  A 100-mm horizontal line is used, with the two extremes of the parameter to be assessed labeled at each end. The patient is asked to indicate their perceived condition by marking a point or drawing a line on the scale that best reflects their current state. VAS is commonly employed to numerically document pain intensity as well as the patient's subjective global health assessment.

SECONDARY OUTCOMES:
Australian Canadian Osteoarthritis Hand Index (AUSCAN) | Patients will be assessed before and after the intervention, and at the 1st and 3rd months following the treatment.
  The AUSCAN Osteoarthritis Hand Index is a validated instrument used to assess the functional status of the hand in individuals with hand osteoarthritis. It evaluates disease-specific health status across three domains: pain (5 items), stiffness (1 item), and physical function (9 items). Patients are asked to report the severity of pain (5 questions; score range: 0-20), stiffness (1 question; score range: 0-4), and functional difficulty (9 questions; score range: 0-36) they have experienced over the past 48 hours. The scale consists of a total of 15 items, with an overall score ranging from 0 to 60. Each item is rated on a 5-point Likert scale: 0 = none, 1 = mild, 2 = moderate, 3 = severe, and 4 = extreme.
Duruöz Hand Index (DHI) | Patients will be assessed before and after the intervention, and at the 1st and 3rd months following the treatment.
  The Duruöz Hand Index (DHI) is a self-administered functional disability questionnaire developed in 1996 specifically for the assessment of hand and wrist function in individuals with rheumatoid hand involvement. It consists of 18 items evaluating daily activities related to hand function, including tasks involving cooking, dressing, personal hygiene, office work, and other general activities. Responses are rated using a Likert scale ranging from 0 to 5 (0 = no difficulty, 5 = impossible to perform). The total score ranges from 0 to 90, with higher scores indicating greater functional impairment. Factor analysis of the DHI has identified a four-dimensional structure: activities requiring grip strength, manual dexterity, finger grip strength, and finger dexterity.
Functional Index of Hand Osteoarthritis (FIHOA) | Patients will be assessed before and after the intervention, and at the 1st and 3rd months following the treatment.
  The Functional Index for Hand Osteoarthritis (FIHOA) is a validated questionnaire consisting of 10 items that reflect daily activities requiring hand use. Each item is scored on a 4-point scale ranging from 0 to 3, where 0 indicates no difficulty, 1 = mild difficulty, 2 = considerable difficulty, and 3 = impossible to perform. The total score ranges from 0 to 30. Lower scores indicate better hand function, whereas higher scores reflect greater functional impairment.
Short Form-36 (SF-36) | Patients will be assessed before and after the intervention, and at the 1st and 3rd months following the treatment.
  The Short Form-36 (SF-36) is a widely used health-related quality of life questionnaire composed of 36 items distributed across eight subscales: physical functioning, role limitations due to physical health, role limitations due to emotional problems, bodily pain, social functioning, mental health, vitality, and general health perceptions. It assesses the individual's health status over the past four weeks. Each subscale is scored, and the responses are transformed into a 0 to 100 scale, with 0 representing the worst possible health status and 100 representing the best. The SF-36 also includes two summary component scores: the Physical Component Summary (PCS) and the Mental Component Summary (MCS). The PCS is derived from the physical functioning, role-physical, bodily pain, and general health subscales, whereas the MCS is composed of the vitality, social functioning, role-emotional, and mental health subscales.
Pinch Strength | Patients will be assessed before and after the intervention, and at the 1st and 3rd months following the treatment.
  Pinch strength will be assessed using a calibrated pinch gauge (Baseline® Hydraulic Pinch Gauge). The measurement will be performed with the patient seated, the shoulder in adduction and neutral rotation, the elbow flexed at 90°, the forearm in a neutral position, and the wrist positioned between 0°-30° of dorsiflexion and 0°-15° of ulnar deviation. To minimize the effects of fatigue, a one-minute rest interval will be provided between each measurement. The test will be repeated three times, and the mean of the three trials will be recorded.
Grip Strength | Patients will be assessed before and after the intervention, and at the 1st and 3rd months following the treatment.
  Grip strength will be measured using a calibrated hydraulic hand dynamometer (Jamar® Hydraulic Hand Dynamometer). Similar to the pinch strength assessment, a one-minute rest interval will be provided between each trial to minimize fatigue. The measurement will be repeated three times, and the average value will be recorded. During the assessment, the patient will be seated with the shoulder in adduction and neutral rotation, the elbow flexed at 90°, the forearm in a neutral position, and the wrist maintained between 0°-30° of dorsiflexion and 0°-15° of ulnar deviation.

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University, Kayseri, Turkey (Türkiye)